CLINICAL TRIAL: NCT03228485
Title: The Feasibility and Acceptability of a (Mobile) Application for Men With LUTS/BPH: a Pilot Study
Brief Title: Benign Prostatic Hyperplasia (BPH) Mobile Application Pilot Study
Status: Completed | Type: Observational
Sponsor: Société Internationale d'Urologie (Other)
Responsible Party: Sponsor
Other Study IDs: uCARE-2018-002
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Smartphone; Application; Pilot; mhealth
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MyBPH Care: All patients enrolled in this study.
  Interventions: Device: MyBPH Care mobile app

INTERVENTIONS:
Device: MyBPH Care mobile app — The application that will give daily medication reminders and via which the questionnaires can be filled out.

SUMMARY:
This study assesses the feasibility, and acceptability of a (mobile) application for men presenting at their physician's office with LUTS/BPH; starting with medical therapy and naïve for treatment. Patients will be enrolled in the study by their physician (GP or urologist). The patients will receive a daily medication reminder including frequent feedback on medication adherence. Furthermore, standard questionnaires will be filled out via the application. The hypothesis of this pilot study is that application is feasible and accepted in this group of patients.

DETAILED DESCRIPTION:
Rationale:

One of the next developments in healthcare is digitalization, including (mobile) applications that could support healthcare providers. A significant number of aging men suffer from lower urinary tract symptoms (LUTS), often caused by benign prostate hyperplasia (BPH). LUTS/BPH is primarily treated by physicians (GPs or Urologists). Optimal evaluation of patients with LUTS/BPH, treatment selection and follow-up by the physicians and medication adherence are essential in the management of LUTS. This pilot project represents a strong collaboration between a urological association, urologists, and physicians in supporting healthcare improvement for LUTS/BPH with the use of a (mobile) application. The hypothesis is that the (mobile) application can support the patient in medication adherence and improve the adherence by feedback and that the application can help to collect objective disease information with electronic questionnaires.

Objectives:

The primary objective is to assess the feasibility, and acceptability of a (mobile) application for men presenting at their general practitioner/or urologist with LUTS/BPH who are either: under treatment, or who may require medical therapy for the first time.

The secondary objectives are to identify potential gaps, clarify controversial points of the application, to document the communication between patients, physicians and supervising urologists in order to optimize (if necessary) the application, to assess medication adherence and to record if treatment provided by physicians is in compliance with the guidelines recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age ≥ 40
* Bothersome LUTS
* Start of medical therapy for LUTS
* Either:

  1. No previous LUTS/BPH treatment (medical or invasive), or
  2. Under medical treatment
* In possession of a smartphone, tablet or computer with internet connection
* Access to email
* Fluent speaking and reading of the national language
* Signed informed consent

Exclusion Criteria:

* Previous LUTS/BPH treatment with surgery
* Previous pelvic surgery or radiotherapy
* History of neurological disease
* History of bladder or prostate cancer
* Unable to provide informed consent
* Analphabet
* Unable to operate a smartphone/ tablet/computer
* Incapable of understanding the language in which the information for the patient is given

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be men, age ≥ 40, presenting at their physician's office with LUTS/BPH symptoms and are either: a) treatment naïve for LUTS/BPH or b) under medical treatment.
  The study will be conducted by five centers in five countries: Institute for Monitoring of Urogenital Diseases in Larissa, Greece, the Istanbul Medipol University in Turkey, the Hospital Universitario la Zarzuela in Spain, the Hospital de San António in Portugal, and the University of Florence in Italy. The participating physicians will be from these areas and thus so will the participants.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of a mobile application for LUTS | 6 months
  The feasibility is assessed by the application use for men presenting at their general practitioner/or urologist with LUTS/BPH who are either: under treatment, or who may require medical therapy for the first time. The patient application will be judged as Definitely Feasible if the study is completed for ≥70% eligible patients, Possibly Feasible (completed for 50-69% eligible patients) or Not Feasible (completed for <50%).

SECONDARY OUTCOMES:
Acceptability and satisfaction of a mobile application for LUTS | 6 months
  In order to assess the acceptance and satisfaction of the mobile application including the application subjective quality and perceived impact, a questionnaire will be used. This questionnaire is based on a standardized application rating questionnaire, namely the user Mobile Application Rating Scale (uMARS). Outcomes are described and compared between centers.
Medication adherence | 6 months
  Self-reported medication adherence by the patient via the application over the full period of the pilot.
Compliance to guidelines | At baseline
  Descriptive comparison between the medication prescribed by the physician and the advised medication according to the international guidelines based on the patient characteristics.
Referral network | At the end of the 6 months period
  Evaluation of the referral communication between the physicians and the supervising urologist by questions in the final questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Gravas, MD, Study Chair — Societe Internationale d'Urologie
Locations (5):
- University Hospital of Larissa, Institute for Monitoring of Urogenital Diseases, Larissa, Greece
- University of Florence, Florence, Italy
- Hospital de Santo Antonio, Porto, Portugal
- Hospital Universitario la Zarzuela, Madrid, Spain
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided